CLINICAL TRIAL: NCT00797485
Title: Maintenance and Reinduction Chemotherapy With Avastin in Metastatic Colon Cancer: The MARTHA (SICOG 0803) Trial
Brief Title: Bevacizumab and Combination Chemotherapy in Treating Patients With Previously Untreated Metastatic Colorectal Cancer That Cannot Be Removed By Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern Italy Cooperative Oncology Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000617983; SICOG-0803; EudraCT-2008-004890-17
Record Dates: First submitted 2008-11-22; First posted 2008-11-25 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-06

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Capecitabine; Fluorouracil; Irinotecan; Leucovorin

ARMS (2):
- Arm I (Active Comparator): Patients receive bevacizumab IV over 30-90 minutes on day 1. Patients also receive FOLFIRI chemotherapy comprising irinotecan hydrochloride IV over 1 hour and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours on days 1 and 2. Treatment repeats every 2 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium
- Arm II (Experimental): Patients receive bevacizumab and FOLFIRI chemotherapy (B-FOLFIRI) as in arm I. Treatment repeats every 2 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive bevacizumab IV over 30-90 minutes on day 1 and oral capecitabine once every 12 hours on days 1-14. Treatment repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: capecitabine; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium

INTERVENTIONS:
Biological: bevacizumab — Given IV
Drug: capecitabine — Given orally
  Arms: Arm II
Drug: fluorouracil — Given IV
Drug: irinotecan hydrochloride — Given IV
Drug: leucovorin calcium — Given IV

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase III trial is studying how well giving induction therapy with bevacizumab together with combination chemotherapy with or without capecitabine followed by bevacizumab maintenance therapy in treating patients with metastatic colorectal cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare two strategies of induction bio-chemotherapy followed by the same maintenance biotherapy in terms of time to failure in patients with previously untreated metastatic colorectal cancer.

Secondary

* To compare the two arms of treatment in terms of response rate, duration of responses, progression-free survival, safety, and quality of life of these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to treatment center, performance status (0 vs 1), and number of metastatic sites (1 vs ≥ 2). Patients are randomized to 1 of 2 induction therapy arms.

* Arm I: Patients receive bevacizumab IV over 30-90 minutes on day 1. Patients also receive FOLFIRI chemotherapy comprising irinotecan hydrochloride IV over 1 hour and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours on days 1 and 2. Treatment repeats every 2 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive bevacizumab and FOLFIRI chemotherapy (B-FOLFIRI) as in arm I. Treatment repeats every 2 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive bevacizumab IV over 30-90 minutes on day 1 and oral capecitabine once every 12 hours on days 1-14. Treatment repeats every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

In both arms, patients achieving stable disease after completion of 6 months of induction therapy proceed to maintenance therapy.

* Maintenance therapy: Patients receive bevacizumab IV over 30-90 minutes every 3 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.

During or after completion of maintenance therapy, patients with tumor regrowth that is not classified as disease progression from baseline and who achieved partial or complete response during or after their induction therapy proceed to reinduction therapy.

* Reinduction therapy: Patients receive B-FOLFIRI as described previously. Quality of life is assessed at baseline, every 3 months during induction therapy, and at discontinuation of study therapy.

After completion of study therapy, patients are followed for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed colorectal cancer

  * Metastatic disease that is not amenable to surgery
* At least one measurable lesion according to RECIST criteria
* No untreated brain metastases or spinal cord compression

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 12 weeks
* Hemoglobin ≥ 9.0 g/dL
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and/or ALT ≤ 2.5 times ULN (< 5 times ULN if liver metastases present)
* Alkaline phosphatase ≤ 2.5 times ULN (< 5 times ULN if liver metastases present)
* PT-INR/PTT < 1.5 times ULN
* Creatinine clearance > 50 mL/min OR serum creatinine ≤ 1.5 times ULN
* Proteinuria on dipstick urinalysis < 2+ OR 24-hour urine protein ≤ 1g
* Not pregnant or nursing
* Negative pregnancy test
* Must be accessible for treatment and follow-up
* No history of inflammatory bowel disease and/or acute or subacute bowel occlusion
* No serious non-healing wound, ulcer, or bone fracture
* No evidence of bleeding diathesis or coagulopathy
* No uncontrolled hypertension
* No clinically significant cardiovascular disease including any of the following:

  * Cerebrovascular accident within the past 6 months
  * Myocardial infarction within the past 6 months
  * Unstable angina
  * New York Heart Association grade II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
* No known allergy to Chinese hamster ovary cell proteins or any of the components of the study medications
* No other malignancy within the past 5 years except basal cell and squamous cell skin cancer or carcinoma in situ of the cervix
* No significant traumatic injury within the past 28 days
* No substance abuse or medical, psychological, or social conditions that may interfere with participation in the study or the evaluation of study results
* Able to swallow oral medications

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 6 months since prior adjuvant treatment
* No prior irinotecan and/or bevacizumab during prior adjuvant therapy
* No prior cytotoxic drugs for the metastatic disease
* More than 10 days since prior and no concurrent anticoagulants for therapeutic purposes
* No chronic, daily treatment with high-dose aspirin (> 325 mg/day) or other medications known to predispose to gastrointestinal ulceration
* No treatment with any investigational drug within the past 30 days
* No major surgical procedure or open biopsy within the past 28 days or anticipated need for a major surgical procedure during the course of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Estimated)
Dates: Start 2008-07; Primary Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Time to failure of strategy

SECONDARY OUTCOMES:
Response according to RECIST criteria
Duration of response
Progression-free survival
Safety according to NCI CTCAE v3.0
Quality of life as assessed by EORTC QLQ-C30 questionnaire (v 3.0) at baseline, every 3 months during induction chemotherapy, and at discontinuation of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Comella, MD, Principal Investigator — Istituto Nazionale per lo Studio e la Cura dei Tumori
Locations (1):
- Southern Italy Cooperative Oncology Group, Naples, Italy